CLINICAL TRIAL: NCT03539861
Title: Immunomodulatory Biomimetic Device to Treat Myocardial Stunning in End-stage Renal Disease Patients (ERSD)
Brief Title: Immunomodulatory Biomimetic Device to Treat Myocardial Stunning in End-stage Renal Disease Patients
Acronym: ESRD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID- pandemic, nursing shortages. enrolled two patients then not enough nurses in dialysis unit to be able to attend to patients
Sponsor: University of Michigan (Other)
Collaborators: Renal Research Institute (Other)
Responsible Party: Principal Investigator, Lenar Yessayan, Associate Professor of Internal Medicine, Medical School, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HUM00125836
Record Dates: First submitted 2018-05-16; First posted 2018-05-29 (Actual); Results first posted 2023-01-17 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2022-11

CONDITIONS: End Stage Renal Disease; Acute Kidney Injury; Chronic Kidney Disease Stage 5
Keywords: End Stage Renal Disease; Hemodialysis; Chronic Kidney Disease Stage 5
MeSH Terms: conditions — Kidney Failure, Chronic; Acute Kidney Injury; Renal Insufficiency, Chronic | interventions — Renal Dialysis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Hemodialysis (Other): The treatment arm (all participants are in this arm) is done in two phases that are described below:
  Treatment 1 will be standard hemodialysis (no device).
  Treatment 2 will be hemodialysis with the study device. Of importance, this 5 hour session is planned to ensure adequate solute clearance but with only 4 hour high ultrafiltration to achieve the patients dry weight.
  Interventions: Device: Hemodialysis

INTERVENTIONS:
Device: Hemodialysis — Each patient will receive two hemodialysis treatments while on this study. The first hemodialysis treatment will be standard of care hemodialysis. The second treatment will be the experimental hemodialysis treatment using the Selective cytopheretic device.
  Other Names: Selective cytopheretic device; SCD; SCD filter anticoagulated with regional citrate

SUMMARY:
Hemodialysis is a therapy that filters waste, removes extra fluid and balances electrolytes. In hemodialysis, blood is removed from the body and filtered through a man-made membrane called a dialyzer, and then the filtered blood is returned to the body. Hemodialysis is associated with injury to the heart muscle called myocardial stunning. This may occur for many reasons, including removal of fluid during dialysis or low blood pressure. Initial ischemia and subsequent white blood cell infiltration into the injured myocardium play a critical role in the degree of myocardial ischemia reperfusion injury.

In this study an additional man made membrane (selective cytopheretic device) and tubing will be added to the dialysis circuit. The device shifts the circulating white blood cells pool to a less inflammatory phenotype. Researchers believe the selective cytopheretic device will alter the phenotype of circulating white blood cells which play a role in myocardial stunning.

The purpose of this study is to evaluate whether the selective cytopheretic device will reduce myocardial stunning events in hemodialysis patients. It will also report the rate of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* End-stage renal disease (Chronic Kidney Disease Stage 5)
* Receiving hemodialysis 3 times/week for over 3 months
* Baseline blood pressure before hemodialysis has been ≥ 100/50 over preceding 4 weeks
* Recurrent weight gain between hemodialysis sessions

Exclusion Criteria:

* Any active inflammatory condition (e.g., gout, systemic lupus erythematosus flare, hepatitis B or C infection, allograft rejection, subcutaneous injection of illicit drugs, "skin popping")
* Treatment with immunosuppressive therapy within 30 days of study
* Blood levels within a specified range
* Woman who is pregnant, breast feeding a child, or is trying to become pregnant
* Heart weakness or failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2021-08-04 (Actual); Study Completion 2021-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lenar Yessayan, Principal Investigator — The University of Michigan Department of Internal Medicine
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Hemodialysis: The treatment arm (all participants are in this arm) is done in two phases that are described below:
  Treatment 1 will be standard hemodialysis (no device).
  Treatment 2 will be hemodialysis with the study device. Of importance, this 5 hour session is planned to ensure adequate solute clearance but with only 4 hour high ultrafiltration to achieve the patients dry weight.
  Hemodialysis: Each patient will receive two hemodialysis treatments while on this study. The first hemodialysis treatment will be standard of care hemodialysis. The second treatment will be the experimental hemodialysis treatment using the Selective cytopheretic device.
Period: Overall Study
Arm/Group | Hemodialysis
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Hemodialysis
Number analyzed (Participants) | 2
Age, Customized [Count of Participants; unit: Participants]
  25-30 | 1
  62-68 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 1
  Black or African-American | 1
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Regional Wall Abnormalities Identified on Echocardiogram
Description: Regional wall motion will be scored using a standard wall motion scoring scheme. (1= normal; 2=hypokinetic; 3= akinetic; 4=dyskinetic). Scores will be tabulated for each of 16 predefined segments and a global wall motion score calculated as the sum of individual scores divided by the number visualized segments.
Time Frame: Baseline, 5 hour, 24 hours
Population: Regional wall motion was not able to be evaluated for one participant because of arrhythmia. Because sharing data about the other individual could violate privacy concerns, it is not analyzed or displayed.
Arm/Group | Hemodialysis
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Participants With an Adverse Event Based on the Clinical Laboratory Measurement: Ionized Calcium (iCa)
Description: Number of participants who experienced a clinically significant change in systemic ionized calcium compared to reference range: 1.12 to 1.30.
Time Frame: Hour 1, hour 2, hour 3, hour 4, hour 5
Measure: Count of Participants; unit: Participants
Arm/Group | Hemodialysis
Number analyzed (Participants) | 2
Participants | 0

3. Secondary Outcome: Number of Participants With an Adverse Event Based on the Clinical Laboratory Measurement: Hemoglobin
Description: Number of participants who experienced a clinically significant change in hemoglobin who experience a change of more than 10% of baseline
Time Frame: Baseline, Hour 5, 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Hemodialysis
Number analyzed (Participants) | 2
Participants | 0

ADVERSE EVENTS:
Time Frame: 8 days
Arm/Group | Hemodialysis
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-26): https://cdn.clinicaltrials.gov/large-docs/61/NCT03539861/Prot_SAP_000.pdf